CLINICAL TRIAL: NCT06719011
Title: A Randomized, Placebo Controlled and Double-blinded Study Assessing the Safety, Tolerability, Pharmacokinetics, and Efficacy of Subcutaneous Administrations of NNC0174 1213 in Male Participants With Overweight or Obesity.
Brief Title: A Study on How NNC0174-1213 Works in People With Overweight or Obesity.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NN9839-8082; U1111-1308-5620 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: NNC0174-1213 (SD1-SD5) (Experimental): Part A: Single ascending dose (SAD) of NNC0174-1213 will be administered in cohorts 1-5.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)
- Part A: Cagrilintide (SDA and SDB) (Experimental): Part A: Single ascending dose (SAD): Cagrilintide SDA will be administered in cohort 1 and 2.
  Cagrilintide SDB will be administered in cohort 3 and 4.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)
- Part A: Placebo (Experimental): Part A: Single ascending dose (SAD) of placebo will be administered to cohorts 1-5.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)
- Part B: NNC0174-1213 (MD1-MD5) (Experimental): Part B: Multiple ascending doses (MAD) of NNC0174-1213 will be administered to cohorts 1-5.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)
- Part B: Cagrilintide (MDA) (Experimental): Part B: Multiple ascending doses (MAD) of Cagrilintide MDA will be administered to cohorts 1-5.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)
- Part B: Placebo (Experimental): Part B: Multiple ascending doses (MAD) of placebo will be administered to cohorts 1-5.
  Interventions: Drug: NNC0174-1213 A; Drug: Cagrilintide B; Drug: Placebo A (NNC0174 1213 A)

INTERVENTIONS:
Drug: NNC0174-1213 A — Participants will be randomized to receive NNC0174-1213 A administered as subcutaneous (s.c. under the skin) injection.
  Single ascending dose (SAD) will be injected for Part A cohorts and multiple ascending doses (MAD) will be injected for Part B cohorts.
Drug: Cagrilintide B — Participants will be randomized to receive Cagrilintide B administered as subcutaneous (s.c. under the skin) injection.
  Single ascending dose (SAD) will be injected for Part A cohorts and multiple ascending doses (MAD) will be injected for Part B cohorts.
Drug: Placebo A (NNC0174 1213 A) — Participants will be randomized to receive Placebo administered as subcutaneous (s.c. under the skin) injection.
  Single ascending dose (SAD) will be injected for Part A cohorts and multiple ascending doses (MAD) will be injected for Part B cohorts.

SUMMARY:
This study is testing a new study medicine to treat people living with overweight or obesity. The aim of this study is to see if the medicine is safe, how it works in human body, and what human body does to the study medicine. Participants will either get the new study medicine NNC0174-1213, a study medicine called "cagrilintide" or a placebo (a "dummy medicine" similar to the new study medicine and study medicine but without active ingredients). Which treatment participants will get is decided by chance. The new study medicine and the study medicine are potential new medicines which cannot be prescribed by doctors. This study will last for about a year in total.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 27.0 and 34.9 kilogram per meter square (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Body weight more than or equal to (>=) 80.0 kilograms (kg) at screening.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Exposure to an investigational medicinal product within 2 months or 5 half-lives of the investigational medicinal product (if known), whichever is longer, before screening.
* Participants report prior receipt of an amylin and/or calcitonin receptor agonist within the last 6 months.
* Impaired liver function defined as any of the below:
* Aspartate aminotransferase (AST) more than or equal to (>=) 2 times upper limit of normal at screening
* Alanine aminotransferase (ALT) more than or equal to (>=) 2 times upper limit of normal at screening
* Bilirubin more than (>) 1.5 times upper limit of normal at screening (except if known or proven Gilbert's syndrome)
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) less than (<) 75 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) at screening.
* Glycated haemoglobin (HbA1c) more than or equal to (>=) 6.5 percent (%) (48 millimoles per mole (mmol/mol) at screening.
* Any clinically significant body weight change more than or equal to (>=) 5 percent (%) self-reported change) or dieting attempts (e.g., participation in a weight reduction program) within 90 days before screening .
* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:
* Vitamin D (25-hydroxycholecalciferol) less than (<) 12 nanogram per milliliter (ng/mL) (30 nanometer (nM) at screening
* Parathyroid hormone (PTH) outside normal range at screening
* Total calcium outside normal range at screening
* Calcitonin more than or equal to (>=) 50 nanogram per liter (ng/L) at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of treatment emergent adverse events (TEAE) reported by participants exposed to NNC0174 1213 | From NNC0174 1213 administration (Day 1) to completion of the end of study visit (Day 46)
  Number of events
Part B: Number of treatment emergent adverse events (TEAE) | From first administration (Day 1) to completion of the end of study visit (Day 67)
  Number of events

SECONDARY OUTCOMES:
Part A: AUC; area under the NNC0174 1213 plasma concentration-time curve | From pre-dose on Day 1 to completion of the end of study visit (Day 46)
  measured in hour*nanomoles per liter (h*nmol/L).
Part A: Cmax; maximum observed NNC0174 1213 plasma concentration | From pre-dose on Day 1 to completion of the end of study visit (Day 46)
  measured in nanomoles per liter (nmol/L).
Part B: AUC; area under the NNC0174 1213 plasma concentration-time curve | From first administration (Day 1) to completion of the end of study visit (Day 67)
  measured in h*nmol/L.
Part B: Cmax; maximum observed NNC0174 1213 plasma concentration | From first administration (Day 1) to completion of the end of study visit (Day 67)
  measured in nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - ICON Early Phase Services, LLC, San Antonio, Texas
  - ICON Early Phase Services, LLC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com